CLINICAL TRIAL: NCT05505071
Title: DANTE SPACE for Evaluation of Subjects With Intracranial Vascular Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution and study will not be started.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-2096
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Vascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DANTE SPACE MRI Sequence (Experimental): Participants will receive an additional DANTE SPACE sequence with their clinical MRI
  Interventions: Device: DANTE SPACE sequence

INTERVENTIONS:
Device: DANTE SPACE sequence — investigational MRI sequence less than 15 minutes
  Other Names: Delay Alternating with Nutation for Tailored Excitation (DANTE)

SUMMARY:
Purpose: The purpose of this study is to evaluate the Delay Alternating with Nutation for Tailored Excitation (DANTE) SPACE sequence in clinical studies to determine whether it can provide more useful information for clinical diagnosis.

Participants: 100 participants with concern for intracranial vascular disease scheduled to undergo a clinical vessel wall MRI will be recruited.

Procedures (methods): Patients with concern for intracranial vascular disease scheduled to undergo a clinical vessel wall MRI who will have an additional non-FDA approved sequence (DANTE SPACE) added to their clinical scan. The investigational sequence requires less than 15 minutes and will be added following the standard MRI sequence.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Concern for intracranial vascular disease
* Scheduled to undergo a clinical vessel wall MRI

Exclusion Criteria:

* Claustrophobia
* Implanted metallic devices, parts, vascular clips, or other foreign bodies.
* Known hypersensitivity to gadolinium contrast or to any component of gadolinium contrast refractory to standard medications (antihistamines, steroids)
* Impaired kidney function (serum creatinine level > 1.8 mg/dL or a glomerular filtration rate < 60 as approximated using serum creatinine levels) unless anuric and on dialysis.
* Any woman who is pregnant or has reason to believe she is pregnant via self report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Utility for Visualizing Pathology | Baseline
  The primary objective is to determine the percent of participants with a visible region of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmud Mossa-Basha, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months after and continuing for 36 months following publication
Access Criteria: The investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.